CLINICAL TRIAL: NCT05607979
Title: The RENEW Study: (Restoring Tissue and Evaluating Novel Treatments for Efficacy in Wounds): A Non-Inferiority Study
Brief Title: Restoring Tissue and Evaluating Novel Treatments for Efficacy in Wounds
Acronym: RENEW
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lavior Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RENEW-01
Record Dates: First submitted 2022-10-29; First posted 2022-11-07 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Foot Ulcer
Keywords: diabetes; diabetic foot ulcer; wound; hydrogel; diabetes mellitus
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized controlled, double-blinded clinical Non-inferiority trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: The Study Participant, The Care Provider, and the Investigator are all blinded from the treatments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TRIAL INTERVENTION (Active Comparator): Trial intervention is wound treatment with Lavior Diabetic Wound Gel.
  Interventions: Drug: Lavior Diabetic Wound Gel
- CONTROL THERAPY (Active Comparator): Control therapy is defined as Smith & Nephew Solosite Gel Hydrogel Wound Dressing, according to actual guidelines or local clinical standards. Standard therapy is defined as the currently accepted and widely used treatment for the respective wound type, based on the results of past research. Therapy options for standard wound care are treatments that experts agree to be appropriate, accepted, and widely used.
  Interventions: Drug: Smith & Nephew Solosite Gel Hydrogel Wound Dressing

INTERVENTIONS:
Drug: Lavior Diabetic Wound Gel — Daily application of hydrogel treatment for 60 days.
  Arms: TRIAL INTERVENTION
Drug: Smith & Nephew Solosite Gel Hydrogel Wound Dressing — Daily application of hydrogel treatment for 60 days.
  Arms: CONTROL THERAPY

SUMMARY:
This is an IRB-approved multicenter study.This non-inferiority study aims to evaluate differential healing rates between Lavior Diabetic Wound Gel and other Hydrogels. Study therapy will be started in the outpatient setting and followed accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Foot Wound in the setting of Diabetes Mellitus
* Written informed consent
* Minimum wound surface area of 0.7 x 0.7 cm (0.49 square cm)

Exclusion Criteria:

* Age < 18 years
* Noncompliance with study procedures, visit schedule or follow up Gangrene and/or untreatable Peripheral Arterial Disease
* Malignancy of the wound
* Use of any other hydrogels not being studied in this investigation within 1 month of being enrolled
* Dry, uninfected, stable pressure ulcers of the heel
* Dry, stable eschar in arterial wounds
* Simultaneous participation in competing clinical trials
* Pregnancy or Nursing mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint | 60 days
  The primary endpoint of this trial is defined as time (number of days) to achieve complete wound closure in study participants where closure was observed on or before Day 60. The primary endpoint of this trial is defined as time (number of days) to achieve complete wound closure in study participants where closure was observed on or before Day 60.

SECONDARY OUTCOMES:
Incidence of wound closures within 60 days | 60 days
  The incidence of wound closure achieved within each treatment arm will be evaluated after a maximum study observation/treatment period of 60 days
Recurrence | 60 days
  Recurrence of wound opening after initial closure and confirmed wound closure will be assessed and compared between the treatment groups.
Change in wound depth over time (cm) | 60 Days
  Change in wound depth (cm) over time will be evaluated by measurement of wound depth (cm) over time
Change in wound surface area over time (cm) | 60 Days
  Change in wound surface area (cm) over time will be evaluated by measurement of wound surface area (cm) over time.
Change of wound size over time (cm) | 60 days
  Change of Necrotic wound bed surface area (cm) will be evaluated by measurement of necrotic area of wound (cm) over time. Photographic details of wound will be captured at each visit with standardized disposable ruler (cm).
Change in Pain Scores over time (60 days) | 60 days
  Change in pain scores will be recorded over time (60 days) through the use of a patient reported 0 -10 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Ho Steve Bae, DPM, Principal Investigator — Baefoot Podiatry
Locations (1):
- Baefoot Podiatry, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No